CLINICAL TRIAL: NCT04619004
Title: HERTHENA-Lung01: A Phase 2 Randomized Open-Label Study of Patritumab Deruxtecan (U3-1402) in Subjects With Previously Treated Metastatic or Locally Advanced EGFR-mutated Non-Small Cell Lung Cancer (NSCLC)
Brief Title: HERTHENA-Lung01: Patritumab Deruxtecan in Subjects With Metastatic or Locally Advanced EGFR-mutated Non-Small Cell Lung Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Collaborators: Daiichi Sankyo Co., Ltd. (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: U31402-A-U201; 2020-000730-17 (EudraCT Number)
Record Dates: First submitted 2020-10-29; First posted 2020-11-06 (Actual); Results first posted 2024-04-02 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Non-Small Cell Lung Cancer Metastatic; Non-Small Cell Lung Cancer With Mutation in Epidermal Growth Factor Receptor
Keywords: Non-Small Cell Lung Cancer Metastatic; Non-Small Cell Lung Cancer with Mutation in Epidermal Growth Factor Receptor; Epidermal growth factor receptor; HER3-DXd; Patritumab Deruxtecan; U3-1402
MeSH Terms: interventions — patritumab deruxtecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Study Group 1: Patritumab deruxtecan 5.6 mg/kg (Experimental): Study Group 1 will be participants with metastatic or locally advanced NSCLC with an EGFR-activating mutation randomized to receive patritumab deruxtecan 5.6 mg/kg IV every 3 weeks (Q3W)
  Interventions: Drug: Patritumab Deruxtecan (Fixed dose)
- Study Group 2: Patritumab deruxtecan Up-Titration (Experimental): Study Group 2 will be participants with metastatic or locally advanced NSCLC with an EGFR-activating mutation randomized to receive patritumab deruxtecan up-titration IV every 3 weeks (Q3W)
  Interventions: Drug: Patritumab Deruxtecan (Up-Titration)

INTERVENTIONS:
Drug: Patritumab Deruxtecan (Fixed dose) — Patritumab deruxtecan will be dosed at 5.6 mg/kg as an intravenous (IV) infusion administered on Day 1 of each 21-day cycle.
  Other Names: U3-1402; HER3-DXd
  Arms: Study Group 1: Patritumab deruxtecan 5.6 mg/kg
Drug: Patritumab Deruxtecan (Up-Titration) — Patritumab deruxtecan will be dosed as an intravenous (IV) infusion administered at Cycle 1, 3.2 mg/kg; Cycle 2, 4.8 mg/kg; Cycle 3 and subsequent cycles, 6.4 mg/kg administered on Day 1 of each 21-day cycle.
  Other Names: U3-1402; HER3-DXd
  Arms: Study Group 2: Patritumab deruxtecan Up-Titration

SUMMARY:
This study is designed to evaluate the antitumor activity of patritumab deruxtecan in participants with metastatic or locally advanced NSCLC with an activating EGFR mutation (exon 19 deletion or L858R) who have received and progressed on or after at least 1 EGFR TKI and 1 platinum-based chemotherapy-containing regimen.

DETAILED DESCRIPTION:
This study will initially randomize participants to one of 2 arms in a 1:1 ratio to receive either a 5.6 mg/kg fixed dose regimen or an up-titration dose regimen of patritumab deruxtecan (HER3-DXd, U3-1402).

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following criteria to be eligible for inclusion in this study.

* Sign and date the tissue informed consent form (ICF) and the main ICF, prior to the start of any study-specific qualification procedures.
* Male or female participants aged ≥18 years (follow local regulatory requirements if the legal age of consent for study participation is >18 years old).
* Histologically or cytologically documented locally advanced or metastatic NSCLC not amenable to curative surgery or radiation.
* Documentation of radiological disease progression while on/after receiving most recent treatment regimen for locally advanced or metastatic disease. Participants must have received both of the following:

  * Prior treatment with osimertinib. Participants receiving an EGFR TKI at the time of signing informed consent should continue to take the EGFR TKI until 5 days prior to Cycle 1 Day 1. Participants in South Korea known to harbor a clinically actionable genomic alteration in addition to EGFR mutation (e.g., anaplastic lymphoma kinase [ALK] or ROS1 protocol oncogene 1 [ROS1] fusion) for which treatment is available must have also received prior treatment with at least 1 approved genotype-directed therapy, unless unable (i.e., if contraindicated). No new testing for these genomic alterations (e.g., ALK or ROS1 fusion) is required for Screening.
  * Systemic therapy with at least 1 platinum-based chemotherapy regimen.
* Documentation of an EGFR-activating mutation detected from tumor tissue or blood sample: exon 19 deletion or L858R.
* At least 1 measurable lesion confirmed by BICR as per RECIST v1.1
* Consented and willing to provide required tumor tissue of sufficient quantity and of adequate tumor tissue content. Required tumor tissue can be provided as either:

  * Pretreatment tumor biopsy from at least 1 lesion not previously irradiated and amenable to core biopsy OR
  * Archival tumor tissue collected from a biopsy performed within 3 months prior to signing of the tissue consent and since progression while on or after treatment with the most recent cancer therapy regimen.
* Eastern Cooperative Oncology Group Performance Standard of 0 or 1 at Screening.
* Has adequate bone marrow reserve and organ function based on local laboratory data within 14 days prior to Cycle 1 Day 1:

  * Platelet count : ≥100,000/mm^3 or ≥100 × 10^9/L (platelet transfusions are not allowed up to 14 days prior to Cycle 1 Day 1 to meet eligibility)
  * Hemoglobin: ≥9.0 g/dL (transfusion and/or growth factor support is allowed)
  * Absolute neutrophil count: ≥1500/mm^3 or ≥1.5 × 10^9/L
  * Serum creatinine (SCr) or creatinine clearance (CrCl): SCr ≤1.5 × upper limit of normal (ULN), OR CrCl ≥30 mL/min as calculated using the Cockcroft-Gault equation or measured CrCl
  * Aspartate aminotransferase/alanine aminotransferase: ≤3 × ULN (if liver metastases are present, ≤5 × ULN)
  * Total bilirubin: ≤1.5 × ULN if no liver metastases (<3 × ULN in the presence of documented Gilbert's syndrome [unconjugated hyperbilirubinemia] or liver metastases)
  * Serum albumin: ≥2.5 g/dL
  * Prothrombin time (PT) or PT-International normalized ratio (INR) and activated partial thromboplastin time (aPTT)/PTT: ≤1.5 × ULN, except for subjects on coumarin-derivative anticoagulants or other similar anticoagulant therapy, who must have PT-INR within therapeutic range as deemed appropriate by the Investigator

Exclusion Criteria:

Participants meeting any exclusion criteria for this study will be excluded from this study.

* Any previous histologic or cytologic evidence of small cell OR combined small cell/non-small cell disease in the archival tumor tissue or pretreatment tumor biopsy.
* Any history of interstitial lung disease (including pulmonary fibrosis or radiation pneumonitis), has current interstitial lung disease (ILD), or is suspected to have such disease by imaging during screening.
* Clinically severe respiratory compromise (based on Investigator's assessment) resulting from intercurrent pulmonary illnesses including, but not limited to:

  * Any underlying pulmonary disorder (eg, pulmonary emboli within 3 months prior to the study enrollment, severe asthma, severe chronic obstructive pulmonary disease [COPD]), restrictive lung disease, pleural effusion);
  * Any autoimmune, connective tissue or inflammatory disorders with pulmonary involvement (eg, rheumatoid arthritis, Sjogren's syndrome, sarcoidosis); OR prior complete pneumonectomy.
* Is receiving chronic systemic corticosteroids dosed at >10 mg prednisone or equivalent anti-inflammatory or any form of immunosuppressive therapy prior to enrollment. Participants who require use of bronchodilators, inhaled or topical steroids, or local steroid injections may be included in the study.
* Evidence of any leptomeningeal disease.
* Evidence of clinically active spinal cord compression or brain metastases.
* Inadequate washout period prior to Cycle 1 Day 1, defined as:

  * Whole brain radiation therapy <14 days or stereotactic brain radiation therapy <7 days;
  * Any cytotoxic chemotherapy, investigational agent or other anticancer drug(s) from a previous cancer treatment regimen or clinical study (other than EGFR TKI), <14 days or 5 half-lives, whichever is longer;
  * Monoclonal antibodies, other than immune checkpoint inhibitors, such as bevacizumab (anti-VEGF) and cetuximab (anti-EGFR) <28 days;
  * Immune checkpoint inhibitor therapy <21 days;
  * Major surgery (excluding placement of vascular access) <28 days;
  * Radiotherapy treatment to more than 30% of the bone marrow or with a wide field of radiation <28 days or palliative radiation therapy <14 days; or
  * Chloroquine or hydroxychloroquine <14 days.
* Prior treatment with an anti-human epidermal growth factor receptor 3 (HER3) antibody or single-agent topoisomerase I inhibitor.
* Prior treatment with an antibody drug conjugate (ADC) that consists of any topoisomerase I inhibitor
* Has unresolved toxicities from previous anticancer therapy, defined as toxicities (other than alopecia) not yet resolved to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) v5.0, Grade ≤1 or baseline. Participants with chronic Grade 2 toxicities may be eligible at the discretion of the Investigator after consultation with the Sponsor Medical Monitor or designee.
* Has history of other active malignancy within 3 years prior to enrollment, except:

  * Adequately treated non-melanoma skin cancer;
  * Superficial bladder tumors (Ta, Tis, T1);
  * Adequately treated intraepithelial carcinoma of the cervix uteri;
  * Low risk non-metastatic prostate cancer (with Gleason score <7, and following local treatment or ongoing active surveillance);
  * Any other curatively treated in situ disease.
* Uncontrolled or significant cardiovascular disease prior to Cycle 1 Day 1
* Active hepatitis B and/or hepatitis C infection, such as those with serologic evidence of viral infection within 28 days of Cycle 1 Day 1.
* Participant with any human immunodeficiency virus (HIV) infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 277 (Actual)
Dates: Start 2021-02-02 (Actual); Primary Completion 2022-11-21 (Actual); Study Completion 2026-01-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Daiichi Sankyo
Locations (123):
- United States (33):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - City of Hope, Duarte, California
  - Moores Cancer Center at the UC San Diego Health, La Jolla, California
  - Pacific Shores Medical Group, Long Beach, California
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - University of California at Irvine, Orange, California
  - Cedars Sinai, West Hollywood, California
  - University of Colorado Denver - Anschutz Medical Campus, Aurora, Colorado
  - Florida Cancer Specialists - South, Fort Myers, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Memorial Healthcare System, Pembroke Pines, Florida
  - Florida Cancer Specialist-North, St. Petersburg, Florida
  - Florida Cancer Specialists-Panhandle, Tallahassee, Florida
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - Florida Cancer Specialists-East, West Palm Beach, Florida
  - Emory University, Dunwoody, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Maryland - Marlene and Stewart Greenebaum Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital (MGH) - Hematology/Oncology, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Harvard Medical School, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Henry Ford Cancer Institute/Henry Ford Hospital, Detroit, Michigan
  - Mount Sinai Hospital, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - Cleveland Clinic - Main Campus, Cleveland, Ohio
  - Providence Portland Medical Center, Portland, Oregon
  - Sarah Cannon Research Institute at Tennessee Oncology - Chattanooga, Chattanooga, Tennessee
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - University of Virginia Cancer Center - Emily Couric Clinical Cancer Center, Charlottesville, Virginia
  - Virginia Cancer Specialist, PC, Fairfax, Virginia
  - University of Washington/Seattle Cancer Care Alliance, Seattle, Washington
- Australia (6):
  - Blacktown Hospital, Blacktown, New South Wales
  - The Chris O'Brien Lifehouse, Camperdown, New South Wales
  - St George Public Hospital, Kogarah, New South Wales
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - St John of God Subiaco Hospital, Subiaco, Western Australia
  - Princess Alexandra Hospital, Woolloongabba
- Karl Landsteiner Institut fÃ¼r Lungenforschung und pneumologische Onkologie c/o Klinik Floridsdorf, Vienna, Austria
- Universitaire Ziekenhuis Gasthuisberg, Leuven, Belgium
- Bulgaria (3):
  - MHAT Uni Hospital OOD, Panagyurishte
  - Complex Oncological Center - Russe, Rousse
  - MHAT Serdika, Sofia
- China (11):
  - Beijing Cancer Hospital, Beijing
  - Jilin Cancer Hospital, Changchun
  - University of Electronic Science & Technology of China (UESTC) - Sichuan Cancer Hospital & Institute (Sichuan Provincial Tumor Hospital, Chengdu
  - Guangdong Academy of Medical Science (GAMS) - Guangdong Provincial Peoples Hospital, Guangzhou
  - The First Affiliated Hospital of College of Medicine Zhejiang University, Hangzhou
  - Harbin Medical University - Tumor Hospital (The Third Affiliated Hospital), Harbin
  - General Hospital of Eastern Theater Command, Nanjing
  - Fudan University - Shanghai Cancer Center FUSCC, Shanghai
  - The First Hospital of China Medical University, Shenyang
  - Union Hospital of Tongji Medical College Huazhong University of Science and Technology, Wuhan
  - Henan Cancer Hospital, Zhengzhou
- France (8):
  - CHU Toulouse - Hopital Larrey, Toulouse, Haute-Garonne
  - University Hospital of Nantes - Thoracic Oncology, Nantes, Loire-Atlantique
  - Centre Leon Berard, Lyon, Rhone
  - Hopital Morvan CHU de Brest, Brest
  - Centre Hospitalier Universitaire de Grenoble, Grenoble
  - Institut Curie, Paris
  - Hopital Pontchaillou, Rennes
  - Gustave Roussy, Villejuif
- Germany (6):
  - Kliniken der Stadt Koeln gGmbH Lungenklinik Merheim, KÃ¶ln, North Rhine-Westphalia
  - Universitaet zu Koeln - Uniklinik Koeln, Cologne, North Rhine-Westphal
  - LungenClinic Grosshansdorf, Großhansdorf, Schleswig-Holstein
  - Universitaet zu Koeln - Uniklinik Koeln, Cologne
  - Kliniken der Stadt Koeln gGmbH Lungenklinik Merheim, Cologne
  - University Cancer Center, Dresden
- Italy (5):
  - Azienda Ospedaliero Universitaria di Parma, Parma, Province Of Parma
  - Azienda Ospedaliero-Universitaria San Luigi Gonzaga, Orbassano, Turin
  - IRCCS - Istituto Scientifico Romagnolo per lo Studio e La Cura Dei Tumori ISRT, Meldola
  - Fondazione IRCCS Istituto Nazionale Tumori, Milan
  - Humanitas Cancer Center, Rozzano
- Japan (15):
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - National Cancer Center Hospital, Tokyo, Chuo-ku
  - National Hospital Organization Shikoku Cancer Center, Matsuyama, Ehime
  - National Hospital Organization Hokkaido Cancer Center, Sapporo, Hokkaido
  - Hyogo Cancer Center, Akashi, Hyōgo
  - National Cancer Center Hospital East, Chiba, Kashiwa-shi
  - The Cancer Institute Hospital of JFCR, Ariake, Koto
  - Sendai Kousei Hospital, Sendai, Miyagi
  - Kansai Medical University Hospital, Hirakata, Osaka
  - Kindai University Hospital, Ōsaka-sayama, Osaka
  - Shizuoka Cancer Center, Sunto-gun, Shizuoka
  - National Cancer Center Hospital, Chuo Ku, Tokyo
  - Niigata Cancer Center Hospital, Chuo Ku Niigata-shi
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
  - National Hospital Organization Hokkaido Cancer Center, Sapporo
- Netherlands Cancer Institute, Amsterdam, Netherlands
- Singapore (3):
  - National University Cancer Institute National University Hospital, Singapore
  - National Cancer Centre Singapore NCCS, Singapore
  - OncoCare Cancer Centre- Gleneagles Medical Centre, Singapore
- South Korea (8):
  - Asan Medical Center, Songpa-gu, Seoul
  - Chungbuk National University Hospital, Cheongju-si
  - Kyungpook National University Chilgok Hospital, Daegu
  - National Cancer Center, Goyang-si
  - Seoul National University Bundang Hospital, Seongnam
  - Seoul National University Hospital, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea, Seoul St. Marys Hospital, Seoul
- Spain (10):
  - Hospital Universitario Virgen Macarena, Seville, Andalusia
  - Catalan Institute of Badalona Hospital Germans Trias i Pujol ICO, Badalona, Cataluã'a
  - Hospital Universitario Puerta de Hierro de Majadahonda, Majadahonda, Madrid
  - Hospital Universitario Vall d'Hebron, Barcelona
  - MD Anderson Cancer Center, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - START Madrid - Hospital Universitario HM Sanchinarro, Madrid
  - Hospital Regional Universitario Carlos Haya, Málaga
  - Hospital Clinico Universitario Lozano Bleza, Zaragoza
- Taiwan (8):
  - National Cheng Kung University Hospital, Tainan, Tai Nan Shi
  - E-Da Hospital, Kaohsiung City
  - Chang Gung Memorial Hospital CGMH - Kaohsiung Branch, Niaosong
  - Taichung Veterans General Hospital, Taichung
  - Chung Shan Medical University Hospital, Taichung
  - National Taiwan University Hospital NTUH, Taipei
  - MacKay Memorial Hospital, Taipei
  - Chang Gung Memorial Hospital - Linkou Branch, Taoyuan District
- United Kingdom (4):
  - University Hospital Birmingham NHS Trust, Birmingham
  - The Royal Marsden NHS Foundation Trust, London
  - University College London Hospitals, London
  - The Christie Hospital, Manchester

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Derived] Yu HA, Goto Y, Hayashi H, Felip E, Chih-Hsin Yang J, Reck M, Yoh K, Lee SH, Paz-Ares L, Besse B, Bironzo P, Kim DW, Johnson ML, Wu YL, John T, Kao S, Kozuki T, Massarelli E, Patel J, Smit E, Reckamp KL, Dong Q, Shrestha P, Fan PD, Patel P, Sporchia A, Sternberg DW, Sellami D, Janne PA. HERTHENA-Lung01, a Phase II Trial of Patritumab Deruxtecan (HER3-DXd) in Epidermal Growth Factor Receptor-Mutated Non-Small-Cell Lung Cancer After Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitor Therapy and Platinum-Based Chemotherapy. J Clin Oncol. 2023 Dec 10;41(35):5363-5375. doi: 10.1200/JCO.23.01476. Epub 2023 Sep 10. PMID 37689979
- [Derived] Yu HA, Yang JC, Hayashi H, Goto Y, Felip E, Reck M, Vigliotti M, Dong Q, Cantero F, Fan PD, Kanai M, Sternberg DW, Janne PA. HERTHENA-Lung01: a phase II study of patritumab deruxtecan (HER3-DXd) in previously treated metastatic EGFR-mutated NSCLC. Future Oncol. 2023 Jun;19(19):1319-1329. doi: 10.2217/fon-2022-1250. Epub 2023 May 22. PMID 37212796

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 277 participants were enrolled and randomized to treatment at clinical sites in the United States, Japan, Republic of Korea, Singapore, Taiwan, Austria, Belgium, Bulgaria, France, Germany, Italy, Netherlands, Spain, United Kingdom, and Australia. Two participants did not receive any treatment. (1 person in each treatment arm).
Groups:
- Patritumab Deruxtecan 5.6 mg/kg: Participants with metastatic or locally advanced NSCLC with an EGFR-activating mutation and who received patritumab deruxtecan 5.6 mg/kg IV every 3 weeks (Q3W)
- Patritumab Deruxtecan Up-Titration: Participants with metastatic or locally advanced NSCLC with an EGFR-activating mutation and who received a patritumab deruxtecan up-titration regimen
Period: Overall Study
Arm/Group | Patritumab Deruxtecan 5.6 mg/kg | Patritumab Deruxtecan Up-Titration
Started | 226 | 51
Completed (Ongoing patients as of data cutoff date) | 87 | 14
Not Completed | 139 | 37
Not completed — Death | 114 | 28
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 24 | 7
Not completed — Other - Not specified | 0 | 1

BASELINE CHARACTERISTICS:
Population: Demographic and baseline characteristics were reported from the Full Analysis Set.
Groups:
- Patritumab Deruxtecan Up-Titration: Participants with metastatic or locally advanced NSCLC with an EGFR-activating mutation and received a patritumab deruxtecan up-titration regimen
- Total: Total of all reporting groups
Arm/Group | Patritumab Deruxtecan 5.6 mg/kg | Patritumab Deruxtecan Up-Titration | Total
Number analyzed (Participants) | 226 | 51 | 277
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.7 (9.86) | 59.8 (10.07) | 62.2 (9.95)
Age, Customized [Count of Participants; unit: Participants]
  <65 years | 122 | 36 | 158
  ≥65 years | 104 | 15 | 119
  <75 years | 201 | 49 | 250
  ≥75 years | 25 | 2 | 27
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 133 | 29 | 162
  Male | 93 | 22 | 115
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 106 | 32 | 138
  Black or African-American | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  White | 92 | 15 | 107
  Other | 24 | 3 | 27

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) as Assessed by Blinded Independent Central Review (BICR)
Description: ORR is defined as the proportion of participants with a best overall response (BOR) of confirmed complete response (CR) or confirmed partial response (PR) as assessed by BICR per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. CR was defined as a disappearance of all target lesions and PR was defined as at least a 30% decrease in the sum of diameters of target lesions based on RECIST v1.1.
Time Frame: Data collected from screening until time of disease progression by BICR, death, lost to follow up, study discontinuation, whichever occurs first, assessed up to approximately 21 months
Population: Objective response rate was assessed in the Efficacy Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Patritumab Deruxtecan 5.6 mg/kg | Patritumab Deruxtecan Up-Titration
Number analyzed (Participants) | 225 | 50
Participants | 64 | 8

2. Secondary Outcome: Duration of Response (DoR)
Description: DoR is defined as the time from the first documented confirmed response (CR or PR) to the date of progression or death due to any cause as assessed by BICR and Investigator per RECIST v1.1, respectively. CR was defined as a disappearance of all target lesions and PR was defined as at least a 30% decrease in the sum of diameters of target lesions.
Time Frame: as for outcome 1
Population: Duration of response rate was assessed in participants with confirmed CR or PR in the Efficacy Analysis Set.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Patritumab Deruxtecan 5.6 mg/kg | Patritumab Deruxtecan Up-Titration
Number analyzed (Participants) | 64 | 8
months
  Duration of response (BICR) | 6.0 [4.4 to 7.2] | 7.1 [2.8 to 15.2]
  Duration of response (Investigator): number analyzed (Participants) | 56 | 8
  Duration of response (Investigator) | 6.9 [5.6 to 7.2] | 5.1 [2.6 to 9.5]

3. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS is defined as the time from the start of study treatment to the first documentation of objective progressive disease (PD) per RECIST v1.1 or death due to any cause. PFS will be determined by BICR and by Investigator, respectively.
Time Frame: as for outcome 1
Population: Progression-free survival was assessed in the Efficacy Analysis Set.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Patritumab Deruxtecan 5.6 mg/kg | Patritumab Deruxtecan Up-Titration
Number analyzed (Participants) | 225 | 50
months
  Progression-free survival (BICR) | 5.5 [5.1 to 5.9] | 6.7 [4.2 to 8.8]
  Progression-free survival (Investigator) | 5.5 [4.2 to 5.7] | 5.3 [4.0 to 8.2]

4. Secondary Outcome: Objective Response Rate (ORR) as Assessed by the Investigator
Description: ORR is defined as the proportion of participants with a BOR of confirmed CR or confirmed PR as assessed by the Investigator per RECIST v1.1. CR was defined as a disappearance of all target lesions and PR was defined as at least a 30% decrease in the sum of diameters of target lesions.
Time Frame: Data collected from screening until time of disease progression, death, lost to follow up, study discontinuation, whichever occurs first, assessed up to approximately 21 months
Population: Objective response rate was assessed in the Efficacy Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Patritumab Deruxtecan 5.6 mg/kg | Patritumab Deruxtecan Up-Titration
Number analyzed (Participants) | 225 | 50
Participants | 56 | 8

5. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR is defined as the proportion of participants who achieved a BOR of confirmed CR, confirmed PR, or stable disease (SD) as assessed by BICR and by the Investigator per RECIST v1.1, respectively. CR was defined as a disappearance of all target lesions, PR was defined as at least a 30% decrease in the sum of diameters of target lesions, and stable disease (SD) was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD; at least a 20% increase in the sum of diameters of target lesions.
Time Frame: as for outcome 1
Population: Disease control rate was assessed in the Efficacy Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Patritumab Deruxtecan 5.6 mg/kg | Patritumab Deruxtecan Up-Titration
Number analyzed (Participants) | 225 | 50
Participants
  Disease control rate (BICR) | 166 | 38
  Disease control rate (Investigator) | 169 | 37

6. Secondary Outcome: Time to Tumor Response (TTR)
Description: TTR is defined as the time from the start of study treatment to the date of the first documentation of confirmed response (CR or PR) as assessed by BICR and Investigator per RECIST v1.1, respectively. CR was defined as a disappearance of all target lesions and PR was defined as at least a 30% decrease in the sum of diameters of target lesions.
Time Frame: as for outcome 1
Population: Time to response rate was assessed in participants with confirmed CR or PR in the Efficacy Analysis Set.
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Patritumab Deruxtecan 5.6 mg/kg | Patritumab Deruxtecan Up-Titration
Number analyzed (Participants) | 64 | 8
months
  Time to response (BICR) | 2.2 (1.31) | 1.7 (0.61)
  Time to response (Investigator): number analyzed (Participants) | 56 | 8
  Time to response (Investigator) | 2.5 (1.78) | 2.1 (1.09)

7. Secondary Outcome: Best Percentage Change in the Sum of Diameters (SoD) of Measurable Tumors
Description: The best percentage change in the SoD of measurable tumors is defined as the percentage change in the smallest SoD from all post-baseline tumor assessments, taking as reference the baseline SoD.
Time Frame: as for outcome 1
Population: Percentage change in the sum of diameters was assessed in participants with available data in the Efficacy Analysis Set.
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | Patritumab Deruxtecan 5.6 mg/kg | Patritumab Deruxtecan Up-Titration
Number analyzed (Participants) | 210 | 49
percentage change from baseline
  Sum of diameters (BICR) | -25.66 (30.39) | -17.48 (29.54)
  Sum of diameters (Investigator): number analyzed (Participants) | 208 | 48
  Sum of diameters (Investigator) | -20.84 (27.01) | -11.46 (29.25)

8. Secondary Outcome: Overall Survival (OS)
Description: OS defined as the time from the start of study treatment to the date of death due to any cause.
Time Frame: Death date is collected until the participant discontinues the study or up to approximately 45 months
Reporting Status: Not Posted, anticipated posting 2025-11

9. Secondary Outcome: Incidence of Treatment Emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs), and Adverse Events of Special Interest (AESIs)
Description: A TEAE is defined as an adverse event (AE) with a start or worsening date during the on-treatment period. A serious AE is defined as any untoward medical occurrence that at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is an important medical event, or may jeopardize the participant or may require medical or surgical intervention to prevent one of the other outcomes noted. AESIs will also be assessed. Adverse events will be coded using MedDRA and will be graded using NCI-CTCAE v5.0.
Time Frame: From baseline up to Day 47 post last dose
Reporting Status: Not Posted, anticipated posting 2025-11

ADVERSE EVENTS:
Time Frame: Adverse events were collected from after first dose up to 47 days post last dose, up to approximately 21 months (primary outcome data cutoff date).
Description: Safety events are reported from the Safety Analysis Set. Treatment-emergent adverse events are reported per the investigator.
Arm/Group | Patritumab Deruxtecan 5.6 mg/kg | Patritumab Deruxtecan Up-Titration
All-Cause Mortality (participants affected / at risk) | 114/225 | 28/50
Serious Adverse Events (participants affected / at risk) | 90/225 | 16/50
Other Adverse Events (participants affected / at risk) | 223/225 | 49/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patritumab Deruxtecan 5.6 mg/kg (N=225) | Patritumab Deruxtecan Up-Titration (N=50)
Disease progression (General disorders) | 11 (11) | 4 (4)
Pyrexia (General disorders) | 3 (3) | 1 (1)
Asthenia (General disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0)
Malaise (General disorders) | 2 (2) | 0 (0)
Non-cardiac chest pain (General disorders) | 2 (2) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 5 (5) | 0 (0)
COVID-19 (Infections and infestations) | 2 (2) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 0 (0)
Septic shock (Infections and infestations) | 2 (2) | 0 (0)
Bacterial sepsis (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Infectious pleural effusion (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 5 (5) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Duodenal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enterocolitis haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatic duct obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 6 (6) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 5 (6) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (4) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 4 (4) | 1 (1)
Aphasia (Nervous system disorders) | 2 (2) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Normal pressure hydrocephalus (Nervous system disorders) | 1 (2) | 0 (0)
Petit mal epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Metastasis to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 2 (2) | 0 (0)
Hepatic cytolysis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic haematoma (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hypertransaminaemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Transfusion reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cardiac tamponade (Cardiac disorders) | 2 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac disorder (Cardiac disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patritumab Deruxtecan 5.6 mg/kg (N=225) | Patritumab Deruxtecan Up-Titration (N=50)
Nausea (Gastrointestinal disorders) | 147 (215) | 32 (48)
Constipation (Gastrointestinal disorders) | 77 (95) | 15 (19)
Diarrhoea (Gastrointestinal disorders) | 62 (91) | 11 (21)
Vomiting (Gastrointestinal disorders) | 60 (70) | 11 (15)
Stomatitis (Gastrointestinal disorders) | 26 (30) | 7 (7)
Abdominal pain (Gastrointestinal disorders) | 19 (20) | 5 (6)
Abdominal pain upper (Gastrointestinal disorders) | 14 (15) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 14 (19) | 2 (6)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 7 (8) | 3 (3)
Fatigue (General disorders) | 69 (79) | 12 (14)
Asthenia (General disorders) | 41 (70) | 7 (14)
Pyrexia (General disorders) | 22 (30) | 6 (8)
Oedema peripheral (General disorders) | 20 (22) | 3 (3)
Malaise (General disorders) | 15 (23) | 6 (16)
Platelet count decreased (Investigations) | 65 (88) | 13 (22)
Neutrophil count decreased (Investigations) | 61 (104) | 15 (32)
White blood cell count decreased (Investigations) | 48 (85) | 9 (20)
Aspartate aminotransferase increased (Investigations) | 38 (56) | 9 (13)
Alanine aminotransferase increased (Investigations) | 26 (39) | 9 (15)
Weight decreased (Investigations) | 23 (24) | 9 (9)
Blood alkaline phosphatase increased (Investigations) | 21 (25) | 1 (1)
Lymphocyte count decreased (Investigations) | 16 (27) | 3 (4)
Blood lactate dehydrogenase increased (Investigations) | 13 (15) | 1 (1)
Blood creatinine increased (Investigations) | 12 (18) | 3 (4)
Decreased appetite (Metabolism and nutrition disorders) | 92 (115) | 21 (28)
Hypokalaemia (Metabolism and nutrition disorders) | 37 (49) | 6 (8)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 20 (27) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 15 (18) | 2 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 15 (18) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 74 (107) | 15 (23)
Thrombocytopenia (Blood and lymphatic system disorders) | 33 (59) | 5 (5)
Neutropenia (Blood and lymphatic system disorders) | 23 (35) | 5 (13)
Leukopenia (Blood and lymphatic system disorders) | 12 (17) | 1 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 57 (57) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 13 (15) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 40 (44) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 37 (40) | 5 (7)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 22 (27) | 1 (2)
Headache (Nervous system disorders) | 26 (28) | 9 (13)
Dysgeusia (Nervous system disorders) | 14 (17) | 1 (1)
Dizziness (Nervous system disorders) | 13 (16) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 21 (25) | 7 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 20 (22) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 7 (7) | 3 (6)
COVID-19 (Infections and infestations) | 20 (23) | 3 (3)
Pneumonia (Infections and infestations) | 11 (12) | 3 (3)
Urinary tract infection (Infections and infestations) | 10 (12) | 3 (3)
Insomnia (Psychiatric disorders) | 17 (17) | 5 (5)
Vision blurred (Eye disorders) | 6 (6) | 4 (4)
Fall (Injury, poisoning and procedural complications) | 6 (7) | 4 (4)
Hypertension (Vascular disorders) | 5 (5) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-31): https://cdn.clinicaltrials.gov/large-docs/04/NCT04619004/Prot_SAP_000.pdf